CLINICAL TRIAL: NCT06930560
Title: HEARS Neuropsychiatric Symptoms & Hearing Loss: Addressing Hearing Loss as a Common Unmet Contributor of Neuropsychiatric Symptoms
Brief Title: HEARS-NPS: Addressing Hearing Loss as a Common Unmet Contributor of Neuropsychiatric Symptoms
Acronym: HEARS-NPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB00357244; 5R01AG076525-02 (NIH)
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease; Dementia; Hearing Loss; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Hearing Loss; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Experimental)
  Interventions: Device: HEARS-NPS device; Behavioral: HEARS-NPS program
- Delayed treatment (Placebo Comparator)
  Interventions: Device: HEARS-NPS device; Behavioral: HEARS-NPS program

INTERVENTIONS:
Device: HEARS-NPS device — Tailored fitting and programming of a personal sound amplifier accompanied by an aural rehabilitation component.
Behavioral: HEARS-NPS program — Tailored aural rehabilitation for participant and care partner.

SUMMARY:
This randomized controlled trial study aims to evaluate a revised hearing care intervention for older adults with Alzheimer's Disease and Related Dementias (ADRD). The community-delivered hearing care intervention utilizes tailored strategies to assess impact on communication, neuropsychiatric symptoms (NPS), and care partner distress.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 - 100 years old
* English-speaking
* Diagnosis of probable Alzheimer's Disease or other related dementia according to the core clinical criteria outlined in the National Institute on Aging (NIA) and Alzheimer's Association Guidelines
* Speech frequency pure tone average (0.5- 4 kHz) >25 db in the better-hearing ear; adult onset hearing loss
* Availability of caregiver/study partner who is 18+ to participate in all study-related visits and who provides care supervision
* Stable (for 2 weeks or longer) dosing of medication (e.g. antidepressants, antipsychotics) for neuropsychiatric symptoms

Exclusion Criteria:

* Current self-reported use of hearing aid or amplification device
* Medical contraindication to use hearing aids ( e.g. draining ears)
* Inability to participate in the 1-month follow up

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Distress as assessed by the Neuropsychiatric Inventory (NPI-Q) | Baseline, 6-week, 3-month, and 6-months post-intervention (immediate group). Baseline, 6-week, 3-month, and 6-months post-baseline (Delayed Group)
  Scoring: Each of the 12 NPI-Q domains contains a survey question that reflects symptoms of that domain. Initial responses to each domain question are "Yes" or "No". If the response to the question is "No", the informant goes to the next question. If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale and the associated impact of the symptom manifestations using a 5-point scale. The NPI-Q provides symptom Severity and Distress ratings for each symptom reported, and total Severity and Distress scores reflecting the sum of individual domain scores. Total NPI-Q severity score is the sum of individual symptom scores, ranges from 0 to 36. Higher score is worse
  SEVERITY of the symptom (how it affects the patient):
  1. = Mild (noticeable, but not a significant change)
  2. = Moderate (significant, but not a dramatic change)
  3. = Severe

SECONDARY OUTCOMES:
Hearing Handicap Inventory for the Elderly (HHIE-S) | Baseline, 6-week, 3-month, and 6-months post-intervention (immediate group). Baseline, 6-week, 3-month, and 6-months post-baseline (Delayed Group)
  Higher scores indicate increased hearing handicap.
  Scoring:
  0-8 suggests no hearing handicap 10-24 suggests mild-moderate hearing handicap 26-40 suggests significant hearing handicap An increase in the score from baseline (a positive number) indicates a worsening in hearing handicap.
Relationship Quality as assessed by the Patient-Caregiver Closeness Scale (CG-CR) | Baseline, 6-week, 3-month, and 6-months post-intervention (immediate group). Baseline, 6-week, 3-month, and 6-months post-baseline (Delayed Group)
  The scale assesses the closeness of the caregiver-care recipient relationship with six items. The total score ranges from 14 to 70. A higher total score reflects a better relationship quality.
International Outcome Inventory for Hearing Aids (IOI-HA) Survey | Baseline, 6-week, 3-month, and 6-months post-intervention (immediate group). Baseline, 6-week, 3-month, and 6-months post-baseline (Delayed Group)
  The hearing inventory survey is used to evaluate the effectiveness of alternative interventions such as assistive devices and communication strategies. The total score ranges from 7-35 where higher scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Oh, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Memory and Alzheimer's Treatment Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No